CLINICAL TRIAL: NCT00961012
Title: Lessening the Big Squeeze: The Effect of the Trunk Release on Interface Pressures of Individuals Seated in a High Fowler's Positions
Brief Title: The Big Squeeze (Lessening the Big Squeeze: The Effect of the Trunk Release on Interface Pressures of Individuals Seated in a High Fowler's Positions)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H09-01370
Record Dates: First submitted 2009-08-14; First posted 2009-08-18 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Elderly
Keywords: Randomized control trial; pressure mapping; High Fowler's position; bed; ventilation; slow vital capacity; older adult population; 65 years and older
MeSH Terms: conditions — Bornholm Eye Disease; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Experimenter A places the subject in the High Fowler's position by raising the foot of the bed to its highest position, 50 degrees, and the head of the bed to its highest position, 60 degrees. Experimenter A sets the timer for 8 minutes as per pressure mapping protocol. For more stable values, a "settling time" of 8 minutes is required to factor in creep of the pressure mapping sensors and mattress. Experimenter A aims the laser beam to the top of the scapulae where the subject's shoulder meets the mattress surface. Experimenter B initiates a FSA file with the subject's number, takes a pressure reading once 8 minutes is up, measures the trunk displacement, obtains spirometry readings as per protocol, and takes a measure of discomfort. Experimenter B leaves the room, Experimenter A sets the timer for 5 minutes and opens the randomization/ allocation envelope.
  Interventions: Procedure: The Big Squeeze
- Control group (No Intervention): Experimenter A reminds the subject to remain immobile.
  For both intervention and control group. After the five-minute period, experimenter A calls experimenter B to return. Experimenter B takes a pressure reading, measures the trunk displacement, obtains spirometry readings, and takes a measure of discomfort.

INTERVENTIONS:
Procedure: The Big Squeeze — Trunk release as per MSIP protocol. Standing at the foot of the bed, facing the subject, Experimenter A grasps both ends of the flat sheet to pull the trunk forward and away from the mattress surface. As the trunk release procedure is performed, Experimenter A checks to verify that the laser beam shines through to the opposite wall to confirm that the shoulders have cleared the mattress.
  Arms: Intervention

SUMMARY:
Older adults with a disability tend to spend greater periods of time in bed each day and often over a mealtime. To make it safe for them to eat in bed, the patient is placed in a high Fowler's position. This means that the head and the foot of the bed are raised to sit the person up.

Sitting up in bed increases pressure over the buttocks which can lead to the development of a pressure ulcer. The purpose of this study is to evaluate the impact of the positional change called "the trunk release" on pressure over the buttocks, on breathing and on comfort.

Primary Hypothesis - Performing the trunk release with an older adult population at low risk for pressure ulcer will result in a 5mmHg decrease in the peak pressure index over the sacral-coccygeal area as measured by the peak pressure index using a Force Sensitive Applications (FSA) Pressure Mapping System.

Secondary Hypotheses - Performing the trunk release with an older adult population at low risk for pressure ulcer will result in:

* Improved ventilation as measured by a 0.5 liter increase in slow vital capacity.
* Greater comfort as measured by a two point change on a horizontal numeric scale with word anchors combined with the Wong-Baker faces scale (Appendix D).
* A four-centimetre displacement of the trunk as it extends up towards the head of the bed.

DETAILED DESCRIPTION:
Two research assistants will conduct the study. Experimenter A assists with recruitment of subjects, sets up the test environment and performs the trunk release. Experimenter B acts as the primary data collector and will be kept blind to the purpose of the study.

The randomized allocation indicates if the subject is in the intervention or control group. Experimenter A sets up the study hospital bed fitted with a visco-elastic foam mattress, a fitted sheet, a flat sheet and the torso pressure-sensing mat. For standardization, the mat is aligned with markers set on the bed frame. Subjects will wear hospital pajamas over undergarments. Experimenter B records height, weight, age and gender. Subject is seated in a chair and is instructed in the spirometry maneuver. Once the subject is comfortable with the maneuver, Experimenter A asks the subject to lie supine with their body centered on the bed and with their hands resting on their abdomen. Experimenter A reminds the subject to remain completely immobile for the duration of data collection. Experimenter B takes a baseline measure of discomfort as per protocol. Experimenter A places the subject in the High Fowler's position by raising the foot of the bed to its highest position, 50 degrees, and the head of the bed to its highest position, 60 degrees. Experimenter A sets the timer for 8 minutes as per pressure mapping protocol. For more stable values, a "settling time" of 8 minutes is required to factor in creep of the pressure mapping sensors and mattress. Experimenter A aims the laser beam to the top of the scapulae where the subject's shoulder meets the mattress surface. Experimenter B initiates a FSA file with the subject's number, takes a pressure reading once 8 minutes is up, measures the trunk displacement, obtains spirometry readings as per protocol, and takes a measure of discomfort. Experimenter B leaves the room, Experimenter A sets the timer for 5 minutes and opens the allocation envelope.

The Principal Investigator will conduct random spot checks to ensure consistency in set-up.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Residents, families, friends and volunteers of Vancouver Community Residential facilities
* Able to understand and follow instructions
* At low risk for bed sores

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Performing trunk release with older adults at low risk for pressure ulcer results in 5mmHg decrease in peak pressure index over the sacral-coccygeal area measured by peak pressure index using Force Sensitive Applications Pressure Mapping System.

SECONDARY OUTCOMES:
Ventilation as measured by a increase or decrease in slow vital capacity. | after 13 minutes of the treatment
Comfort as measured by a horizontal numeric scale with word anchors combined with the Wong-Baker faces scale (Appendix D). | after 13 minutes of the treatment
A displacement of the trunk as it extends up towards the head of the bed. | after 13 minutes of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guylaine Desharnais, Principal Investigator — Vancouver Coastal Health; William C. Miller, Study Director — University of British Columbia; Jeanette A. Boily, Study Director — Vancouver Coastal Health; Pat Camp, Study Director — Vancouver Coastal Health
Locations (4):
- Canada (4):
  - Vancouver General Hospital - Banfield Pavilion, Vancouver, British Columbia
  - George Pearson Centre, Vancouver, British Columbia
  - Dogwood Lodge, Vancouver, British Columbia
  - University of British Columbia Hospital - Purdy Pavilion, Vancouver, British Columbia